CLINICAL TRIAL: NCT02679976
Title: Marketed Contact Lens Real World Through Focus Curve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5728
Record Dates: First submitted 2016-01-22; First posted 2016-02-11 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-07

CONDITIONS: Visual Acuity

ARMS (1):
- Study Lens (etafilcon A) for Multifocal (Experimental): All Subjects in this study will wear the same contact lenses. However subjects wil be stratified as Hyperopes or Myopes using a 1:1 allocation. The study lens will be worn for a period of approximately 4 hours to allow lenses to settle on the eyes.
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: etafilcon A — Marketed Multifocal Contact Lens

SUMMARY:
This is a single-visit prospective study to establish a real world Marketed Contact Lens 'Through Focus Curve' (TFC) measurement by comparing the consistency of vision between myopes and hyperopes. 33 subjects will be enrolled (at least 15 myopes and 15 hyperopes), who are 40 years of age or older, for a 1-visit, 4-hour study for measurements to be taken.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be ≥40 years of age.
* The subjects' optimal vertexed spherical equivalent distance correction must be between -6.00 Diopters (D) and +4.00 D in each eye.
* The subject's refractive cylinder must be ≤ -0.75 D in each eye.
* The subject's ADD power must be in the range of +0.75 to +2.50 D in each eye.
* The subject must have best corrected visual acuity of 20/25 or better for each eye.
* The subject can be either a new contact lens wearer or an existing soft contact lens wearer.

Exclusion Criteria:

* Currently pregnant or lactating.
* Any ocular or systemic allergies that contraindicate contact lens wear.
* Any ocular or systemic disease, autoimmune disease, or use of medication that contraindicates contact lens wear.
* Any ocular abnormality that may interfere with contact lens wear.
* Use of any ocular medication, with the exception of rewetting drops.
* Any previous intraocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, and conjunctival injection) which may contraindicate contact lens wear.
* History of herpetic keratitis.
* Any ocular infection or inflammation.
* Any corneal distortion or irregular cornea.
* History of binocular vision abnormality or strabismus.
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV).
* History of diabetes.
* Participant in unrelated research involving test product within 30 days before planned study visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Optometry Technology Group, Ltd., London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 30 subjects were enrolled into this study. Subjects were stratified as either Hyperope or Myopes using a 1:1 allocation. All enrolled subjects completed the study.
Groups:
- Etafilcon A (Multi-focal): All subjects wore etafilcon A(multi-focal) during the study. Subjects were stratified as either Myopes or Hyperopes based on their sphere power.
Period: Overall Study
Arm/Group | Etafilcon A (Multi-focal)
Started | 30
Hyperopes | 16
Myopes | 14
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Arm/Group | Etafilcon A (Multi-focal)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2
  American Indian Or Alaska Native | 0
  Black or African American | 16
  Native Hawaiian or Other Pacific Islander | 0
  White | 10
  Other | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30

OUTCOME MEASURES:

1. Primary Outcome: Distance Binocular LogMAR Visual Acuity
Description: Distance Binocular LogMAR Visual Acuity was measured at 4m for Low luminance ( 2.5 CD/M^2 ), Medium luminance ( 50 CD/M^2 ) and High luminance ( 250 CD/M^2 )
Time Frame: 4 Hr. Post Fitting
Population: The analysis population includes all subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: -10*LogMAR
Groups:
- Etafilcon A (Multi-focal)- Hyperopes; Etafilcon A (Multi-focal)- Myopes: All subjects wore etafilcon A(multi-focal) during the study. Subjects were stratified as either Myopes or Hyperopes based on their sphere power.
Arm/Group | Etafilcon A (Multi-focal)- Hyperopes | Etafilcon A (Multi-focal)- Myopes
Number analyzed (Participants) | 16 | 14
-10*LogMAR
  Low Luminance; N=16, N=14 | -1.072 (0.8748) | -0.904 (1.1423)
  Medium Luminance; N=16, N=14 | 0.9017 (0.450) | 0.557 (0.9465)
  High Luminance; N=16, N=14 | 1.488 (0.6960) | 1.471 (1.650)

2. Primary Outcome: Near Binocular LogMAR Visual Acuity
Description: Near Binocular LogMAR Visual Acuity was measured at 40cm for Low luminance ( 2.5 CD/M^2 ), Medium luminance ( 50 CD/M^2 ) and High luminance ( 250 CD/M^2 )
Time Frame: 4 Hr. Post Fitting
Population: The analysis population includes all subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: -10*LogMAR
Arm/Group | Etafilcon A (Multi-focal)- Hyperopes | Etafilcon A (Multi-focal)- Myopes
Number analyzed (Participants) | 16 | 14
-10*LogMAR
  Low Luminance; N=16, N=14 | -2.278 (1.6989) | -2.261 (1.7030)
  Medium Luminance; N=16, N=14 | -0.591 (1.4003) | -0.650 (1.5274)
  High Luminance; N=16, N=14 | 0.828 (0.9910) | 0.786 (1.0480)

3. Primary Outcome: Intermediate Binocular LogMAR Visual Acuity
Description: intermediate Binocular LogMAR Visual Acuity was measured at 67cm for Low luminance ( 2.5 CD/M^2 ), Medium luminance ( 50 CD/M^2 ) and High luminance ( 250 CD/M^2 )
Time Frame: 4 Hr. Post Fitting
Population: The analysis population includes all subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: -10*LogMAR
Arm/Group | Etafilcon A (Multi-focal)- Hyperopes | Etafilcon A (Multi-focal)- Myopes
Number analyzed (Participants) | 16 | 14
-10*LogMAR
  Low Luminance; N=16, N=14 | -1.544 (1.0355) | -1.318 (1.4770)
  Medium Luminance; N=16, N=14 | -0.075 (0.8367) | 0.043 (1.1410)
  High Luminance; N=16, N=14 | 1.056 (0.7616) | 1.157 (0.7037)

ADVERSE EVENTS:
Arm/Group | Etafilcon A (Multi-focal)
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days